CLINICAL TRIAL: NCT02147899
Title: A Phase 2, Multi-center, Prospective, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effectiveness and Safety of SYM-1219 for the Treatment of Women With Bacterial Vaginosis
Brief Title: A Phase 2 Study of SYM-1219 to Treat Bacterial Vaginosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Symbiomix Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYM-1219-201
Record Dates: First submitted 2014-05-16; First posted 2014-05-28 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — secnidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SYM-1219 Low Dose (Experimental): Administered orally
  Interventions: Drug: SYM-1219
- SYM-1219 High Dose (Experimental): Administered orally
  Interventions: Drug: SYM-1219
- Placebo (Placebo Comparator): Administered orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYM-1219 — Oral
  Other Names: Secnidazole
  Arms: SYM-1219 High Dose; SYM-1219 Low Dose
Drug: Placebo — Oral
  Arms: Placebo

SUMMARY:
The purpose of this research study is to test the safety and effectiveness of the oral investigational new drug, SYM-1219, for the treatment of bacterial vaginosis.

DETAILED DESCRIPTION:
:This was a Phase 2, multi-center, prospective, randomized, double-blind, placebo-controlled study to evaluate the effectivenessand safety of SYM-1219 in women with bacterial vaginosis. Patients determined to be eligible for the study were randomized to one of the following treatments: SYM-1219 1 gram orallyas a single dose;SYM-1219 2 grams orally as a single dose;or matching placebo. Patients determined to be eligible based on the clinical assessments at the Baseline visit (Day 1) were randomized in a 1:1:1 ratio and received a singledose of the assigned study treatment on Day 1 under fasted conditions (i.e., no food 2 hours prior to or 1 hour after dosing). The centralized randomization was stratified by the number of reported episodes of BV in the past 12 months (including the current episode): 3 or fewer episodes versus 4 or more episodes. Patients were asked to complete a daily telephone questionnaire on Days1to7 and at the Test of Cure (TOC)/End of Study (EOS)visit. Patients were also contacted by telephone once on Day 8 to 10 to inquire about possible adverse events (AEs). A TOC visit was conducted between Day 21 and 30; or at EOSif the final visit was notconducted between Day 21and30

ELIGIBILITY:
Inclusion Criteria:

* Are females at least 18 years of age in good general health who are not menopausal.
* Have a clinical diagnosis of bacterial vaginosis, defined as having all of the following criteria:
* Off-white (milky or gray), thin, homogeneous vaginal discharge
* Vaginal pH ≥ 4.7
* Presence of clue cells of ≥ 20% of the total epithelial cells on microscopic examination of the vaginal saline wet mount
* A positive 10% KOH Whiff test.
* Have a Gram stain slide Nugent score ≥ 4 at the Baseline visit (Day 1)

Exclusion Criteria:

* Are pregnant, lactating, or planning to become pregnant during the study.
* Are suspected clinically (or confirmed diagnostically) of having alternative causes of vaginal symptoms including candidiasis, Chlamydia trachomatis, Trichomonas vaginalis, Neisseria gonorrhoeae or Herpes simplex.
* Have received antifungal or antimicrobial therapy (systemic or intravaginal) within 14 days prior to the Baseline visit (Day 1).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2014-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Women's Health Care Research Corp., San Diego, California
  - Women's Medical Research Group, LLC, Clearwater, Florida
  - Healthcare Clinical Data, Inc., North Miami, Florida
  - Atlanta North Gynecology, P.C, Roswell, Georgia
  - Wayne State University, Detroit, Michigan
  - Saginaw Valley Medical Research Group, LLC, Saginaw, Michigan
  - Lawrence OB-GYN Clinical Research, LLC, Lawrenceville, New Jersey
  - Scott Eder MD, Plainsboro, New Jersey
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Clinical Research of Philadelphia, LLC, Philadelphia, Pennsylvania
  - The Jackson Clinic, PA, Jackson, Tennessee
  - TMC Life Research, Inc., Houston, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Tidewater Physicians for Women, Virginia Beach, Virginia
  - University of Washington, Harborview Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Hillier SL, Nyirjesy P, Waldbaum AS, Schwebke JR, Morgan FG, Adetoro NA, Braun CJ. Secnidazole Treatment of Bacterial Vaginosis: A Randomized Controlled Trial. Obstet Gynecol. 2017 Aug;130(2):379-386. doi: 10.1097/AOG.0000000000002135. PMID 28697102

RESULTS

PARTICIPANT FLOW:
Groups:
- SYM-1219 Low Dose; SYM-1219 High Dose: Administered orally
  SYM-1219
- Placebo: Administered orally
  Placebo
Period: Overall Study
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
Started | 71 | 72 | 72
Completed | 71 | 72 | 72
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo | Total
Number analyzed (Participants) | 71 | 72 | 72 | 215
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 71 | 72 | 72 | 215
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 72 | 72 | 215
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 8 | 23
  Not Hispanic or Latino | 64 | 64 | 64 | 192
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 71 | 72 | 72 | 215

OUTCOME MEASURES:

1. Primary Outcome: Cure of Bacterial Vaginosis
Description: Clinical Cure is a composite endpoint determined by normalization of the vaginal discharge and a negative KOH "Whiff" test and Clue cells less than 20% of the total epithelial cells on microscopic examination of the vaginal wet mount. (Number of subjects with clinical cure at TOC/EOS)
Time Frame: Study Days 21-30
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
Number analyzed (Participants) | 64 | 62 | 62
Participants
  Clinical Outcome Responder | 33 | 42 | 11
  Non-Responder | 31 | 20 | 51

2. Secondary Outcome: Cure of Bacterial Vaginosis
Description: Number of subjects with therapeutic cure at Test of Cure (TOC)/End of Study (EOS) (clinical cure + normalization of Nugent score)
Time Frame: Study Days 21-30
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
Number analyzed (Participants) | 64 | 62 | 62
Participants | 64 | 62 | 62

3. Secondary Outcome: Number of Patients With Therapeutic Cure
Description: Clinical Cure and Normalization of the Nugent score. The Nugent score is based on a microscopic assessment of a Gram stain of the vaginal fluid.
Time Frame: Study Days 21-30
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
Number analyzed (Participants) | 64 | 62 | 62
Participants | 14 | 25 | 4

4. Secondary Outcome: Number of Patients With a Normal Nugent Score
Description: The Nugent score is determined by a microscopic assessment of a Gram stain of vaginal fluid.
Time Frame: Study Days 21-30
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
Number analyzed (Participants) | 64 | 62 | 62
Participants
  Nugent Score 0-3 (Normal) | 15 | 25 | 4
  Nugent Score ≥4 (Abnormal) | 49 | 37 | 58

ADVERSE EVENTS:
Arm/Group | SYM-1219 Low Dose | SYM-1219 High Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/71 | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 9/71 | 14/72 | 7/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SYM-1219 Low Dose (N=71) | SYM-1219 High Dose (N=72) | Placebo (N=72)
headache (Nervous system disorders) | 1 | 1 | 0
dizziness (Nervous system disorders) | 0 | 1 | 0
dysgeusia (Nervous system disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal odor (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal pruritis (Reproductive system and breast disorders) | 0 | 1 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
ALT increased (Investigations) | 0 | 1 | 0
AST increased (Investigations) | 0 | 1 | 0
Desmoid tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1
Candida (Infections and infestations) | 1 | 0 | 0
Chlamydia (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 1
Gonorrhea (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Vaginal mycosis (Infections and infestations) | 0 | 2 | 1
Tooth abscess (Infections and infestations) | 0 | 1 | 1
Tooth infection (Infections and infestations) | 0 | 1 | 0
Upper respiratory (Infections and infestations) | 0 | 2 | 2
Acute sinusitis (Infections and infestations) | 0 | 0 | 1
Vaginal candidiasis (Infections and infestations) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No